CLINICAL TRIAL: NCT00852228
Title: Optimal Control of Liver Metastases With Intravenous Cetuximab and Hepatic Artery Infusion of Three-drug Chemotherapy in Patients With Liver-only Metastases From Colorectal Cancer. A European Multicenter Phase II Trial
Brief Title: Optimal Control of Liver Metastases From Colorectal Cancer With Cetuximab and Hepatic Artery Infusion of Chemotherapy
Acronym: OPTILIV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Association pour la Recherche sur le Temps Biologique et la Chronothérapie (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other); Merck Serono International SA (Industry); Pfizer (Industry); CRESGE (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPTILIV07; EUDRACT number: 2007-004632-24
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Metastatic Colorectal Cancer; Liver Metastases; Hepatic Lesions
Keywords: colorectal cancer; unresectable metastases; neo-adjuvant chemotherapy; liver metastases; chronotherapy; cetuximab; irinotecan; oxaliplatin; 5-fluorouracil; hepatic artery infusion; Unresectable hepatic lesions; 1 to 3 prior chemotherapy regimens
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chronomodulated HAI chemotherapy (Experimental)
  Interventions: Drug: IV cetuximab; Drug: HAI chronomodulated chemotherapy
- conventional HAI chemotherapy (Experimental)
  Interventions: Drug: IV cetuximab; Drug: HAI conventional chemotherapy

INTERVENTIONS:
Drug: IV cetuximab — Cetuximab is administered every two weeks at the dose of 500 mg/m² over 2h30 (150 minutes).
  Other Names: Erbitux
Drug: HAI chronomodulated chemotherapy — Irinotecan (180 mg/m²) on day 2 as a 6 hour infusion, starting at 2:00, with a peak at 5:00
  Oxaliplatin (85 mg/m²) in split daily doses for 3 days, starting on day 2. Daily sinusoidal infusion duration will last from 10:15 to 21:45, with peak delivery rate at 16:00.
  5-Fluorouracil (2800 mg/m²) in split daily doses for 3 days, alternating with oxaliplatin infusions, starting on day 2. Daily sinusoidal infusions will last from 22:15 to 9:45 , with peak delivery at 4:00.
  Treatments will be repeated every 2 weeks.
  Other Names: Campto; Eloxatin
  Arms: chronomodulated HAI chemotherapy
Drug: HAI conventional chemotherapy — Irinotecan (180 mg/m²) on day 1 as a one hour infusion, then
  Oxaliplatin (85 mg/m²) on day 1 as a two hour infusion, then
  5-Fluorouracil (2800 mg/m²) as a 48 h infusion starting on day 2, after completion of oxaliplatin delivery.
  Treatments will be repeated every 2 weeks.
  Other Names: Campto; Eloxatin
  Arms: conventional HAI chemotherapy

SUMMARY:
The primary objective of the study is to increase by 15% the complete macroscopic resection rate of predominantly liver metastases from metastatic colorectal cancer through combining systemic cetuximab and hepatic artery infusion of three-drug chemotherapy (irinotecan, oxaliplatin and 5-fluorouracil).

DETAILED DESCRIPTION:
Primary end-point: incidence of complete macroscopic resections of liver metastases (R0+R1).

Secondary end-points:

* the rate of histologic complete responses,
* the individual rates of R0 and R1 resections,
* the rate and site(s) of relapse in the resected patients throughout the 3-year span that follows hepatectomy,,
* the relapse-free survival curve and median in the resected patients,
* the progression-free and the overall survival in the patients receiving at least 4 full courses of HAI therapy and in all the patients (intent to treat),
* the objective response rate,
* the rate of adverse events,
* the dose intensities over 3, 6 and 9 courses,
* the per-operative and post-operative complications associated to liver surgery.

The study also includes a pharmacokinetic analysis, a translational research and a rest/activity monitoring investigation.

Open, label, European, non randomized, multicenter, phase II study of intravenous cetuximab (ERBITUX®) and hepatic artery infusion of three-drug chemotherapy (irinotecan, 5-fluorouracil and oxaliplatin) using conventional or chronomodulated delivery (according to institution experience) in patients with liver metastases from colorectal cancer.

Patients undergo partial hepatectomy after 6 ± 3 courses of therapy whenever possible. The minimum of 3 and the maximum of 9 courses before liver surgery depend upon results from iterative onco-surgical evaluations. A minimum of 6 and up to 9 additional courses of therapy will be administered after surgery, depending upon results of liver surgery, pathology report and patient's status. Overall, the patients will receive 9 to 18 courses of protocol therapy.

The interval between the last course of cetuximab-HAI chemotherapy and surgery will be 2 to 4 weeks. Post operative treatment will be initiated 2 to 4 weeks after liver surgery.

TRANSLATIONAL RESEARCH:

1. Pharmacokinetics:

   For a subset of 16 patients (8 on conventional administration and 8 on chronotherapeutic delivery), plasma pharmacokinetics of irinotecan, 5-FU and oxaliplatin and main metabolites will be evaluated after the first course.
2. Rest-Activity monitoring:

   Rest-activity will be monitored with a wrist-worn actigraph (Ambulatory Monitoring, USA) for 1 week prior to treatment onset and during the 2 weeks following treatment onset (3 weeks). This evaluation will be repeated before, during and after the 4th treatment course and before during and after 7th treatment course. Participation of the centers to this investigation will be left optional.

   Time series will be analyzed before, during and after chemotherapy course, with the time courses of the following parameters:
   * Autocorrelation coefficient at 24 h (r24)
   * Dichotomy index I<O
   * Wavelet-based model function at baseline, and deviation from this model function during and after treatment course delivery.
3. Predictive molecular factors:

In primary tumor and/or in metastases obtained any time prior to inclusion and in resected metastases and non tumoral liver:

* EGFR immunohistochemistry and gene expression or amplification and polymorphism.
* K-ras mutations.
* Clock genes polymorphism or mRNA or protein expression.
* Gene polymorphisms or expression for main pharmacology determinants of irinotecan, 5- FU and oxaliplatin efficacy.
* Inflammatory and immune cell subsets infiltration. Whenever possible, a biopsy of a liver metastasis will also be obtained before treatment onset for documenting these translational endpoints.

In serum, upon inclusion and after 3 courses:

· Determination of serum levels of TGFa, EGF, VEGF, IL-6, IL-8, amphiregulin and epiregulin.

In blood cells upon inclusion:

· Constitutive polymorphisms for ADCC (FCII and FCIII), circadian clock and EGFR.

STATISTICAL METHODS AND SAMPLE SIZE:

The main endpoint will be the incidence of macroscopically complete resections of liver metastases (R0+R1). The confidence intervals (CI) for the response rate will be based on the exact binomial distribution.

For the secondary endpoints, rate of histologic complete responses, rate of R0 resections, rate of R1 resections, rate of relapses, rate of objective responses, the results will be estimated with CI based on the exact binomial distribution. Overall survival time (OS) and progression free survival (PFS) will be analyzed by Kaplan Meier curve. Multivariate analysis will be performed using the Cox proportional hazard model. This analysis will include the following factors: center, performance status, gender, liver disease characteristics, leucocyte count and alkaline phosphatases upon inclusion and treatment delivery schedule, Relapse incidence (RI) is defined as the probability of having had a relapse before time t. Death without experiencing a relapse is a competing event. The method of analysis will be therefore the estimation of Cumulative Incidence curve in a competing risk setting. Multivariate analysis will be performed by the Fine & Gray model. All patients achieving complete remission will be analyzed.

The goal is to increase the rate of complete resections (R0+R1) by 15%, i.e. from 15% (p0=0.15) to 30% (p1=0.30). According to the exact single-stage phase II design method, the trial for accepting that p1 is to be preferred to p0 (with a=5% and b=20%) requires 48 patients assessable for response. To obtain 48 patients assessable for response, 60 patients will be included in the trial.

A major additional effect expected further from this combined treatment modality is the increase of complete histologic responses, a secondary endpoint in this trial, from 5% (with systemic chemotherapy) to 20% with combined cetuximab and 3-drug HAI. This improvement should further reduce the risk of relapse in the liver or outside the liver by 15 %, i.e. from 80% to 65%.

Therefore, the total number of patients will be 60 patients, including 48 assessable and 12 estimated as unassessable for technical reasons (i.e. HAI catheter dysfunction within the first 2 months).

ELIGIBILITY:
* Histologically or cytologically confirmed carcinoma of the colon and/or rectum with evidence of liver metastases (new confirmation of metastatic disease is required in case the time interval from last histological diagnosis to enrolment exceeds 3 years).
* Patient with wild type (WT) KRAS tumor status
* Patient whose liver metastases are considered to be non resectable with curative intent in medico-surgical staff meeting. In particular patients with at least one of the following criteria, which prevent complete local treatment of liver metastasis with surgery alone or surgery plus radiofrequency ablation because:

  * less than 30% estimated residual liver after resection
  * disease in contact with liver main vessels
  * documented progressive disease on imaging documents or doubling of serum levels of carcino-embryonic antigen (CEA) or CA19.9 over the past 90 days or less
* Patient with up to three resectable extrahepatic nodules of <= 10 mm
* One, two or three prior chemotherapy lines for colorectal cancer.
* Written informed consent.
* Age >=18 years.
* Patient must be able to comply with the protocol.
* Life expectancy of at least 3 months.
* At least one measurable metastatic liver lesion (as per RECIST criteria).
* World Health Organization performance status of 0 or 1.
* Adequate hematological function: absolute neutrophil count (ANC) >=1.0 x 10^9/L; platelets >=75 x 10^9/L, hemoglobin (Hb) >=8.5 g/dL.
* International normalized ratio (INR) <=1.5 and activated partial thromboplastin time (aPTT) <=1.5 x upper limit of normal (ULN) within 7 days prior to starting study treatment, in the absence of anticoagulant therapy.
* Liver function: serum bilirubin <=1.5 x ULN; alkaline phosphatase and transaminases <5 x ULN (liver metastases).
* Serum creatinine <= 1.5 x ULN.
* Fertile women and men of childbearing potential (<2 years after last menstruation in women) must use effective means of contraception (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile).

Exclusion Criteria:

* Patient whose primary tumor or metastasis displays mutation of K-Ras (codon 12 and/or 13).
* Unresectable extrahepatic diseases.
* More than three resectable extrahepatic nodules.
* Size of extra hepatic nodules > 1 cm
* Prior HAI of the 3 drugs.
* More than 2 prior surgical attempts for metastatic disease
* Prior radiotherapy for metastatic disease
* Known documented intolerance or hypersensitivity to any of the drugs used.
* Sensory neuropathy grade 3 (National Cancer Institute-Common Terminology Criteria for Adverse Events -NCI-CTCAE, Version 3.0).
* Past or current history (within the last 2 years prior to treatment start) of malignancy other than colorectal cancer (patients with curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible).
* Serious, non healing wound, ulcer, or bone fracture.
* Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that puts the patient at high risk for treatment-related complications.
* Pregnancy or lactation
* Fertile women (< 2 years after last menstruation) and men of childbearing potential not willing to use effective means of contraception.

Prior systemic administration of cetuximab or other anti-EGFR agent is not an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-07; Primary Completion 2012-03 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of complete macroscopic resections (R0+R1) of unresectable liver metastases following chemotherapy. | evaluation every 6th week up to 18 weeks

SECONDARY OUTCOMES:
The rate and site(s) of relapse in the resected patients throughout the 3-year span that follows hepatectomy | every 2 month up to 3 years
The relapse-free survival in the resected patients | every 2nd month up to 3 years
The progression-free and the overall survival in the patients receiving at least 4 full courses of HAI therapy and in all the patients (intent to treat) | every 2nd month up to 3 years
The objective response rate | every 6 weeks up to 18 weeks
The rate of adverse events | continuous up to 30 days following end of treatment
The per-operative and post-operative complications associated to liver surgery | continuous up to 3 months following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Francis A. Lévi, M.D., Ph.D., Principal Investigator — Paul Brousse Hospital, Villejuif, France
Locations (14):
- Clinique Saint-Joseph, Liège, Belgium
- France (9):
  - CHU de Bordeaux, Hôpital Saint-André, Bordeaux
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Centre Jean Perrin, Clermont-Ferrand
  - CHRU de Lille, Hôpital Claude Huriez, Lille
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - CHU Toulouse, Toulouse
  - Chronotherapy Unit, Medical Oncology Department, Paul Brousse Hospital, Villejuif
  - Institut Gustave Roussy, Villejuif
- Italy (3):
  - Università G. d'Annunzio, Chieti
  - Azienda Ospedaliera S.Maria Degli Angeli, Pordenone
  - Istituto Regina Elena, Roma
- Hospital Fernando Fonesca, Amadora, Portugal

REFERENCES:
- [Derived] Bouchahda M, Boige V, Smith D, Karaboue A, Ducreux M, Hebbar M, Lepere C, Focan C, Guimbaud R, Innominato P, Awad S, Carvalho C, Tumolo S, Truant S, De Baere T, Castaing D, Rougier P, Morere JF, Taieb J, Adam R, Levi F; ARTBC International. Early tumour response as a survival predictor in previously- treated patients receiving triplet hepatic artery infusion and intravenous cetuximab for unresectable liver metastases from wild-type KRAS colorectal cancer. Eur J Cancer. 2016 Nov;68:163-172. doi: 10.1016/j.ejca.2016.09.011. Epub 2016 Oct 18. PMID 27768923
- [Derived] Levi FA, Boige V, Hebbar M, Smith D, Lepere C, Focan C, Karaboue A, Guimbaud R, Carvalho C, Tumolo S, Innominato P, Ajavon Y, Truant S, Castaing D, De Baere T, Kunstlinger F, Bouchahda M, Afshar M, Rougier P, Adam R, Ducreux M; Association Internationale pour Recherche sur Temps Biologique et Chronotherapie (ARTBC International). Conversion to resection of liver metastases from colorectal cancer with hepatic artery infusion of combined chemotherapy and systemic cetuximab in multicenter trial OPTILIV. Ann Oncol. 2016 Feb;27(2):267-74. doi: 10.1093/annonc/mdv548. Epub 2015 Nov 16. PMID 26578731